CLINICAL TRIAL: NCT04509661
Title: Efficacy and Safety of Inhaled Bronchodilator in Non-cystic Fibrosis Bronchiectasis Patients With Airflow Limitation: a Multicenter, Open-label Randomized Controlled Trial
Brief Title: Efficacy and Safety of Inhaled Bronchodilator in Non-CF Bronchiectasis With Airflow Limitation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Chief of Department of Pulmonary and Critical Care Medicine, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200413
Record Dates: First submitted 2020-04-22; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-04

CONDITIONS: Bronchiectasis Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Indacaterol-Glycopyrronium (110ug/50ug QD inhalation) for one year.
  Interventions: Drug: LABA/LAMA or Placebo inhalation
- Control group (Placebo Comparator): Placebo treatment for the airway limitation.
  Interventions: Drug: LABA/LAMA or Placebo inhalation

INTERVENTIONS:
Drug: LABA/LAMA or Placebo inhalation — Inhaled LABA/LAMA for one year.
  Other Names: Inhaled dual Bronchodilator

SUMMARY:
Airflow limitation is common exist in idiopathic bronchiectasis patients. However, there are few evidence on the treatment of bronchodilator in bronchiectasis with airflow limitation. The efficacy and safety of dual bronchodilator in idiopathic bronchiectasis with airflow limitation are still unclear. Thus, the investigators conduct a multicenter, open-label randomized controlled trial to investigate the efficacy and safety of dual bronchodilator in idiopathic bronchiectasis with airflow limitation.

DETAILED DESCRIPTION:
Airflow limitation is common exist in idiopathic bronchiectasis patients. Our previous studies showed that FEV1<50% is one of the major risk factors for poor prognosis and high incidence of acute exacerbation in patients with bronchiectasis. However, there are few evidence on the treatment of bronchodilator in bronchiectasis with airflow limitation, and there is no recommendation in bronchiectasis guidelines. Moreover, because of the high risk of infection and bacterial colonization in bronchiectasis, there is still unclear whether inhaled corticosteroids or bronchodilators affect the parameters of bronchiectasis. Thus, there is urgent need to optimize the treatment of bronchiectasis with airflow limitation.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic bronchiectasis with FEV1/FVC < 70%

Exclusion Criteria:

* With Asthma
* α-1 antitrypsin deficiency
* Turculosis
* Lung cancer
* Sarcoidosis
* Idiopathic pulmonary fibrosis
* Primary pulmonary hypertension
* Uncontrolled sleep apnea
* Bronchiectasis accepted long-term low dose macrolides
* Pulmonary surgery within 6 months
* Lower respiratory tract infections require antibiotic treatment in 6 weeks
* Upper respiratory tract infection did not recover for at least 7 days
* With Glaucoma or severe prostate hyperplasia that can not use Indacaterol
* Patients allergic to experimental drugs
* Women pregnant, breast-feeding or who planned a pregnancy during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Actue exacerbation | One year
  Times of acute exacerbation

SECONDARY OUTCOMES:
modified Medical Research Council score | Six months
  modified Medical Research Council score for the degree of dyspnea. The minimum value is 0 and maximum value is 4. Higher scores mean a worse outcome.
Leicester Cough Questionnaire | Six months
  Cough Questionnaire for the degree of cough. The minimum value is 1 and maximum value is 21. Higher scores mean a better outcome.
Questionnaire of life-Bronchiectasis | Six months
  Including eight scales: respiratory symptoms; physical, role, emotional, and social functioning; vitality; health perceptions; and treatment burden. For each scale, scores are standardized on a 0-to-100-point scale; higher scores indicate better health-related quality of life.
FEV1, FVC | Six months
  Forced Expiratory Volume In 1s and Forced Vital Capacity.
FEV1% | Six months
  The percent of predicted Forced Expiratory Volume In 1s
Incidence of atrial fibrillation | Six months
  One of common adverse events
Incidence of coronary artery disease | Six months
  One of common adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jin-fu Xu, MD, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China